CLINICAL TRIAL: NCT07001124
Title: Comparative Efficacy of Duochrome Test Verse +1 Blur Test in Detecting Refracting Error Across Different Ages
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/821
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- duochrome test and +1 blur test (Group1) 18-35 (Experimental)
  Interventions: Diagnostic Test: duochrome test and +1 blur test
- duochrome test and +1 blur test (Group1) 36-60 (Active Comparator)
  Interventions: Diagnostic Test: duochrome test and +1 blur test

INTERVENTIONS:
Diagnostic Test: duochrome test and +1 blur test — The participant is seated at a standard testing distance (typically 6 meters or 20 feet). A duochrome chart with black letters on a split red-green background is presented.
  After determining the subjective refraction, a +1.00 diopter (DS) lens is added to the final prescription. The participant is asked to read the distance visual acuity (VA) chart. The expectation is that the visual acuity should drop to 4 lines on Snellen chart (6/24) when the +1.00 DS lens is added. If VA reduces to 6/24: Indicates that the refraction is not over-minused or over-plussed (proper end point of refraction). If VA remains better than 6/24: Suggests the patient was still accommodating, possibly leading to over-minus (in myopes) or under-plus (in hyperopes) and the refraction should be re-evaluated.

SUMMARY:
The comparative efficacy of the duochrome test versus +1 blur test in detecting refractive errors across different ages remains under-explored in current ophthalmic research. While the duochrome test is widely used to refine prescriptions, its standalone effectiveness compared to +1 blur test based refraction has not been thoroughly investigated.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy, accuracy, and reliability of the duochrome test in identifying refractive errors, including myopia and hyperopia across various ages. Refractive errors, including myopia, hyperopia, and astigmatism, are leading causes of visual impairment, requiring precise diagnostic tools. The duochrome test utilizes chromatic aberration to refine prescriptions, whereas the +1 blur test assesses spherical correction accuracy. Despite their clinical use, direct comparative studies remain limited. A total of 33 participants with estimated 10% dropout randomly assigned to undergo both tests. Groups will be based on different ages, Group A (18-35 years)and group B (36-60 years) ..both test (Duochrome test and +1 blur test) will apply on every patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years old.
* Both genders.
* Those who have refractive error.
* Patients with no history of prior eye surgery.
* No active eye diseases affecting visual acuity, such as cataracts or retinal disorders.
* Ability to cooperate with both the duochrome test and +1 blur test.

Exclusion Criteria:

* Patients with severe visual impairment or neurological conditions affecting vision.
* Patients with nystagmus or conditions that could interfere with reliable testing.
* Age below 18 year and above 60 year excluded
* Those patients who don't show their consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Function Index (VF-14) Questionnaire: | 12 Months
  Scores on all activities that the person performed or did not perform because of vision were then averaged, yielding a value from 0 to 4. This value was multiplied by 25, giving a final score from 0 to 100. A score of 100 indicates able to do all applicable activities score of 0 indicates unable to do all applicable activities because of vision
+1 blur test | 12 Months
  Adding a +1.00 diopter (DS) lens to a patient's final refraction and measuring their distance visual acuity (VA). There are 4 questions with 5 different options ranging from 0-4. minimum score is 0 and maximum score is 16 with spherical correction.
Duochrome Test | 12 Months
  A duochrome test chart .There are 4 questions with 5 different options ranging from 0-4. minimum score is 0 and maximum score is 16 with spherical correction.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye professionals clinic (14-S DHA Phase 2 Ghazi road), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No